CLINICAL TRIAL: NCT06333561
Title: Efficacy of HAIC Combined With Lenvatinib and PD-1 Inhibitor in Infiltrative Hepatocellular Carcinoma: an Observational, Real-world Study
Brief Title: HAIC Combined With Lenvatinib and PD-1 Inhibitor in Infiltrative Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, Clinical Professor, Sun Yat-sen University
Other Study IDs: Liver Project 7
Record Dates: First submitted 2024-03-21; First posted 2024-03-27 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma; Lenvatinib; PD-1 Inhibitor; Hepatic Arterial Infusion Chemotherapy
Keywords: Hepatic arterial infusion chemotherapy; Tislelizumab; Toripalimab; Sintilimab; Camrelizumab; Lenvatinib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; tislelizumab; toripalimab; sintilimab; camrelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HAIC+Len+PD-1 inhibitor group: HAIC combined with Lenatinib and PD-1 inhibitor group
  Interventions: Procedure: Hepatic arterial infusion chemotherapy; Drug: Lenvatinib; Drug: Tislelizumab; Drug: Toripalimab; Drug: Sintilimab; Drug: Camrelizumab
- Len group: Lenvatinib alone
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Procedure: Hepatic arterial infusion chemotherapy — Hepatic arterial infusion chemotherapy (HAIC) procedure was performed with FOLFOX regimen: 85 or 135 mg/m2 oxaliplatin from hour 0 to 2 on day 1400 mg/m2 leucovorin from hour 2 to 4 on day 1, and 400 mg/m2 fluorouracil bolus at hour 5 on the day 1; and 2400 mg/m2 fluorouracil over 46 h on days 1 and 2.
  Groups: HAIC+Len+PD-1 inhibitor group
Drug: Lenvatinib — 12 mg (body weight ≥60 kg) , 8 mg (body weight <60 kg) orally once a day
Drug: Tislelizumab — 200mg intravenously every 3 weeks
  Groups: HAIC+Len+PD-1 inhibitor group
Drug: Toripalimab — 240mg intravenously every 3 weeks
  Groups: HAIC+Len+PD-1 inhibitor group
Drug: Sintilimab — 200mg intravenously every 3 weeks
  Groups: HAIC+Len+PD-1 inhibitor group
Drug: Camrelizumab — 200mg intravenously every 3 weeks
  Groups: HAIC+Len+PD-1 inhibitor group

SUMMARY:
Hepatic arterial infusion chemotherapy (HAIC) plus lenvatinib and programmed cell death protein-1 (PD-1) inhibitor have shown promising results for advanced hepatocellular carcinoma (HCC). However, the evidence for infiltrative is limited. In this study, we aimed to describe the efficacy and safety of lenvatinib and PD-1 inhibitor with HAIC plus lenvatinib for infiltrative HCC.

DETAILED DESCRIPTION:
This study is a multicenter, observational real-world study to explore the efficacy, safety of lenvatinib and PD-1 inhibitor with HAIC in advanced infiltrative hepatocellular carcinoma. This study focused on the management of locoregional therapy combined with lenvatinib and PD-1 inhibitor. This study will create a database that will provide clinical parameters and outcomes of patients undergoing HIAC combined lenvatinib and PD-1 inhibitor as standard of care in hopes of answering key clinical questions.

ELIGIBILITY:
Inclusion Criteria:

1. primary infiltrative HCC according to MRI or CT imaging characteristics.
2. Child-Pugh class A or B, and Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
3. Lenvatinib as initial treatment.
4. patients received HAIC and PD-1 inhibitor in HAIC+Len+PD-1 group, patients received Lenvatinib alone in Len group.
5. no history of other malignancies.
6. no tumor thrombus in the atrium or vena cava.

Exclusion Criteria:

1. HCC with tumor capsule.
2. under 18 years or over 75 years.
3. TACE as initial treatment.
4. sorafenib or other systemic therapy with or without PD-1 inhibitor following HAIC.
5. incomplete tumor imaging data.
6. lost to follow-up after treatment within three months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a multicenter, observational real-world study to explore the efficacy, safety of lenvatinib and PD-1 inhibitor with HAIC in advanced infiltrative hepatocellular carcinoma. This study focused on the management of locoregional therapy combined with lenvatinib and PD-1 inhibitor. This study will create a database that will provide clinical parameters and outcomes of patients undergoing HIAC combined lenvatinib and PD-1 inhibitor as standard of care in hopes of answering key clinical questions.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 24 months
  OS is the length of time from the date of inclusion until death from any cause.

SECONDARY OUTCOMES:
Progression-Free-Survival | 12 months
  Progression was defined as progressive disease by independent radiologic review

OTHER OUTCOMES:
Objective response rate | 6 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as the proportion of all included patients whose best overall response (BOR) is either a complete response or partial response.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Duan, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General hospital, Beijing, Beijing Municipality, China